CLINICAL TRIAL: NCT02518178
Title: Khushi Baby (KB): Efficacy and Impact Assessment of Novel Mobile Health Solution for Vaccination Record Keeping in Rural Udaipur, Rajasthan, India
Brief Title: Khushi Baby (KB): Novel Mobile Health Solution for Vaccination Record Keeping in India
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Khushi Baby Inc. (Other)
Collaborators: Indian Institute of Health Management Research (IIHMR) (Unknown); Seva Mandir, India (Unknown); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109440
Record Dates: First submitted 2015-08-01; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: DTP Vaccine Series Completion
Keywords: NFC; randomization; RCT; mHealth; maternal and child health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NFC Sticker (Active Comparator): Participants will receive an NFC (Near Field Communication) sticker, placed on their existing immunization (MAMTA) card. This will serve as a comparator to the NFC necklace while still allowing for patient data to be digitized and utilized by the health service provider, Seva Mandir.
  Interventions: Device: NFC Sticker
- NFC Necklace (Experimental): Participants will receive a necklace with an NFC pendant, which interfaces with the Khushi Baby mobile application to digitize the data. This arm will allow for the assessment of peer influence effects of the necklace as a social symbol.
  Interventions: Device: NFC Necklace
- NFC Necklace + Voice Reminder (Experimental): In addition to the NFC necklace, mothers of the participants in this arm will receive dialect-specific voice call reminders, informing them about the next camp and the importance of vaccinations.
  Interventions: Device: NFC Necklace; Device: Voice Reminder

INTERVENTIONS:
Device: NFC Necklace
  Other Names: Khushi Baby Necklace; Khushi Baby Pendant
  Arms: NFC Necklace; NFC Necklace + Voice Reminder
Device: Voice Reminder — Dialect-specific reminders will be issued to the mother's cell phone, informing about the upcoming immunization camp and the importance of vaccination
  Other Names: Voice Call Reminder; Voice Message
  Arms: NFC Necklace + Voice Reminder
Device: NFC Sticker — NFC Sticker on existing immunization card (MAMTA card) serves as a comparator to the pendant and pendant+voice call arms.
  Arms: NFC Sticker

SUMMARY:
This is a three arm cluster randomized controlled trial where the unit of randomization is the immunization camp. Immunization camps are the sole provider of vaccinations in our study area and have catchment areas of several villages. The 96 immunization camps will be randomized evenly to one of three arms:

1. control arm; where near field communication (NFC) stickers will be placed on existing immunization booklets. These stickers can be scanned using a mobile phone with an installed application whereby information can be entered onto the phone and then scanned onto the sticker
2. pendant only; where the same NFC technology will be placed into a pendant that is worn by the infant, and
3. pendant as described above with voice reminders sent 15 days, 1 day prior, and the day of the scheduled immunization camp dates.

DETAILED DESCRIPTION:
Routine immunization (RI) is an important tool to achieve the UN Millennium Development Goal (MDG) 4 of reducing child mortality by ensuring childhood protection from infectious disease. Recent 2013 estimates found that of approximately 6.3 million children died before their fifth birthday, with 51.8% (3.3 million) of these deaths attributed to infectious diseases (Liu et al., 2014). In regards to vaccine preventable diseases (VPDs), pneumonia (935,000 deaths) and diarrhea (578,000 deaths) were responsible for the most deaths. Measles, pertussis, tetanus, and meningitis, four other vaccine preventable diseases, were responsible for 362,000 deaths in children under five years old. (Liu et al., 2014)

Vaccination is one of the most cost-effective interventions for increasing childhood survival. (WHO, 2009). Global estimates find that current immunization programs save over 2.5 million lives a year (WHO, 2009). Despite the lifesaving potential of vaccines, in 2012 approximately 17% of children, or about 23 million infants, did not receive all the scheduled vaccines (CDC, 2013) and if they were immunized, they often received the vaccinations late (Clark & Sanderson, 2009).

In 1985, the Government of India launched the Universal Immunization Programme (UIP) to protect all infants (0-12 months) against six preventable diseases: tuberculosis, diphtheria, pertussis, tetanus, poliomyelitis, and measles. The goal of UIP was to ensure 100% coverage of all eligible children with one dose of BCG, three doses of DTP and OPV, and one dose of the measles vaccine. According to the Coverage Evaluation Survey (CES) 2009, a nationwide survey covering all States and Union Territories of India conducted during November 2009 to January 2010 by UNICEF, the national fully immunized coverage (FIC) against the six vaccines included in UIP in the age-group of 12-23 month old children was just 61% (CES, 2009). Coverage with third dose of diphtheria, tetanus and pertussis vaccine (DTP3) is a widely accepted global indicator for RI program performance (Lim SS, et al. 2008). India national estimates found DTP3 coverage was 72% (WHO India 2011), against a global target of 90%. The District Level Health Survey 3 (DLHS 3) findings suggest that the retention rate of childhood immunization was in maximum decline between the second round of DT and polio - 70 % and the third round - 56 % (Shekhar & Yadav, 2013).

The proposed study site, the Udaipur district of Rajasthan, has traditionally had lower immunization estimates than national levels while also performing poorly in other key developmental indicators: infant mortality rate (IMR) is 47 per 1000 live births (SRS Bulletin, 2014, GoI) and maternal mortality rate (MMR) is 244 per 100,000 women of reproductive age (MMR Bulletin, 2013).

To counter the long-standing deficiencies in immunization coverage and other health outcomes, a non-governmental organization (NGO) named Seva Mandir began operations in the area starting in 2004. Seva Mandir, has had a long standing relationship with over 700 villages in Rajasthan, with 105 villages participating in their immunization program. Immunization camps take place at regular, expected intervals throughout the month so caregivers are aware of when the scheduled camps will take place. This study area and its partners have conducted a seminal randomized controlled trial on non-monetary incentives to improve immunization coverage (Banerjee A, et al., 2010).

Although there has been a renewed global focus on improving immunization coverage levels (Alonso PL, et al., 2013; Berkley S, et al., 2013), Rajasthan district still performs poorly in routine immunization delivery and reporting. In efforts to improve the delivery and reporting of immunizations, with subsequent gains in proportions of infants fully vaccinated, we will conduct a cluster RCT that employs novel mHealth technologies to improve the reporting of immunization records and to increase the demand for immunizations through the use of voice message reminders.

One of these novel mHealth technologies is the use of a wearable electronic immunization record. This technology couples a mobile application (app) for health workers with a wearable digital pendant (necklace) for individuals that store their updated medical history. The pendant contains a read/writable NFC chip which allows health workers to digitally update a participant's vaccination records with the tap of a phone, and without the need to be connected to a central database. This technology can also be placed into a sticker that could be attached to an immunization booklet which would simplify record keeping. Importantly, this technology can be distinguished from other mHealth solutions as it does not require a centralized database of patients to look up patient specific records. Rather, the solution is decentralized allowing patients to wear their vaccine history on a necklace that can be accessed digitally in the last mile at the point of care. This work extends the use NFC trackers to simply identify patients and count disease occurrence (Marcus, et al., 2009) to medical record storage at the point of care. The potential for the necklace to play a symbolic role for the promotion of health benefits is an additional reason for the chosen form factor.

The pendant with NFC technology was developed by students at Yale as part of a class project and is called "Khushi Baby" (KB). Yale investigators visited the proposed study site to informally solicit local opinions on the proposed pendant and to receive feedback from Seva Mandir immunization teams to make the KB app user friendly. Importantly, this pendant is contextually relevant as many children in this study area wear similar talismans with the local thought being that they promote good health and can prevent coughs

Others have found that the color and shape of insecticide bed nets was a relevant factor in influencing people's willingness-to-buy the ITNs and thereby adopt the intervention in Southern Ethiopia (Gebresilassie & Mariam, 2011). The KB necklace, a unique feature of the system, also merits a deeper investigation into the characteristics that influence its adoption and whether it can generate a peer effect throughout the community which impacts vaccination adherence rates.

In addition to potentially being able to increase demand for vaccination, the NFC chip pendant could potentially improve the quantity and quality of immunization services available through a more efficient monitoring and outreach system. The current paper system is prone to loss of records due to wear and tear over the 9 to 12 month process to complete immunizations. Paper systems also have the disadvantages of being difficult to query, not individually specific as data is aggregated and transferred, and out-dated due to the time lag in data entry. The system to digitize vaccine records makes individually specific data available to remote monitors in real time so that they can better manage: vaccine stock, resource mobilization for camps, and camp reminder messages via automated voice reminders to child's household mobile phones. It also holds promise in improving workflow in the field. Simply scanning the chip quickly brings a child's records and their due vaccines for the visit without guesswork based on otherwise incomplete records. Finally, new information such as events of vaccine denial and reasons for vaccine denials can be automatically recorded to reveal greater insights on the true vaccine demand for a given village.

Data do not only have the potential to inform the service delivery NGO, but in this system, to also connect back with the community being served via voice call reminders. Many mHealth pilots on "push" based reminders systems have shown promise in improving health outcomes in developing countries (e.g. MedicMobile, M-Power, Frontline SMS, Mobile Alliance for Maternal Action); however further evidence must be collected to determine whether personalized voice calls can specifically reduce immunization drop out. An automated backend allows our push system to reach mothers/primary caregivers in villages before their baby is due for his/her next vaccine.

Our approach stands to be successful for several reasons:

* mHealth solutions have been successfully used to improve the quality and efficiency of data collection across a range of health outcomes, even in developing world settings.
* SMS reminders have shown some success to improve immunization coverage and timeliness in other developing areas (Bangure et al., 2015); we look to seek enhancement of this effect through personalized voice reminders in local language.
* Mobile phone ownership and access levels are at an all-time global high. Globally, the number of people owning mobile phones grew from 1 billion in 2000 to 6 billion in 2012 (World Bank, 2012). Reaching the last mile may be facilitated through remote reminder systems that alleviate the burden of local workers hired to go door-to-door, walking tens of miles the day before an immunization camp
* Monthly immunization camps are the predominant avenue for infants to be vaccinated. This immunization delivery system benefits the proposed study as study staff will not have to travel to many different clinics and/or households to track enrolled infant's immunization status.

ELIGIBILITY:
Inclusion Criteria:

* Mother/ Primary Caregiver has an infant between the age of 42 days (minimum age for DTP1 administration per WHO guidelines) and 6 months of age; there is no age restriction for inclusion. In the very rare instance that a male is the primary caregiver, they will also be invited to participate in the study. Survey questions are not gender or age specific, but wil require the caregiver to answer questions about his/her children, socioeconomic and health status, and vaccine awareness.
* Self-identified resident within one of the villages associated with the immunization camp
* Willing to give informed consent (sign or thumbprint)

Exclusion Criteria:

* Infant has received at least 1 dose of DTP vaccine
* Caregiver and infant intends to move before the next 6 camps have been completed (in the next 6-9 months)

Ages: 42 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
20% increase in DTP3 coverage | 6 camps after DTP1 receipt (6 months)
  Comparing necklace (with or without voice call reminders) to control arm infants

SECONDARY OUTCOMES:
Increase in DTP3 coverage for necklace + voice reminder arm compared to other 2 arms | 6 camps after DTP1 receipt (6 months)
Improved camp attendance rates | Over 6 camp period after DTP1 receipt (6 months)
  Comparing camps randomized to receive necklace (with or without voice reminders) to control arm infants.
Retention of pendant compared to that of NFC stickered MAMTA card | 6 camps after DTP1 receipt (6 months)
Increased time efficiency of NFC system (both stickers and pendants) compared to existing paper-based system of recording immunization | Paper log books (status quo control) will be used to establish a baseline for timeliness during first 2 months of the study. In the latter 2 months, the KB app digitization will be timed.
  The surveyor will categorize the times separately for new and follow-up patients. The analysis will consider average times for new registrants and follow up registrants in KB app vs. logbook for each health worker (GNM). These indicators will be used to compile a composite measure of time efficiency.
Increased accuracy between NFC system (both stickers and pendants) compared to existing paper-based system of recording immunization | In the first 2 months, the logbook records will be digitized and de-identified for each camp. In the latter 2 months, the digitization of records will take place exclusively through the KB app.
  At the end of each camp the number of child-specific syringes and complete vaccine vials will be counted by the Surveyor; these will serve as the gold standards. The analysis will examine the frequency of underreporting and overreporting of total vaccines (as determined by syringes) and of individual vaccines (as determined by complete vaccine vials when available); rates of underreporting and overreporting will be examined at the camp level (n=2 for each camp) and after clubbing all camps per month (n= 2 months). These indicators will be used to compile a composite accuracy outcome measure.
Survey-based outcomes: user satisfaction, socio-demographic profile of infants, vaccine awareness of mothers and the differential effects on vaccination adherence | Intake survey at enrollment + follow-up surveys at each camp (approximately once a month during follow-up period)
Failure rate of the Khushi Baby mobile application | Throughout study period of 9 months
  time series data to be collected from the app itself (error logs and internal counters for each replacement); number of entries in backup logbook will be digitized and added

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Shahnawaz, PhD cand, Principal Investigator — Indian Institute of Health Management Research (IIHMR)

REFERENCES:
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870
- [Background] WHO, UNICEF, World Bank. State of the world's vaccines and immunization. 3rd edition. Geneva: World Health Organization; 2009.
- [Background] Clark A, Sanderson C. Timing of children's vaccinations in 45 low-income and middle-income countries: an analysis of survey data. Lancet. 2009 May 2;373(9674):1543-9. doi: 10.1016/S0140-6736(09)60317-2. Epub 2009 Mar 19. PMID 19303633
- [Background] Centers for Disease Control and Prevention (CDC). Global routine vaccination coverage--2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 1;62(43):858-61. PMID 24172880
- [Background] Lim SS, Stein DB, Charrow A, Murray CJ. Tracking progress towards universal childhood immunisation and the impact of global initiatives: a systematic analysis of three-dose diphtheria, tetanus, and pertussis immunisation coverage. Lancet. 2008 Dec 13;372(9655):2031-46. doi: 10.1016/S0140-6736(08)61869-3. PMID 19070738
- [Background] Coverage Evaluation Survey India 2009
- [Background] District Level Health Survey Round 3, 2008-09 India.
- [Background] Annual Health Survey 2012-13 Fact Sheet: Rajasthan. Rajasthan Ministry of Health.
- [Background] Shekhar, C. & Yadav, D. India's Universal Immunisation Programme to prevent children from preventable disease: retention and dropout approach. The Lancet. 2013; 381: S151.
- [Background] Alonso PL, de Quadros CA, Robert M, Lal AA. Decade of Vaccines. Editorial. Vaccine. 2013 Apr 18;31 Suppl 2:B3-4. doi: 10.1016/j.vaccine.2013.02.035. No abstract available. PMID 23598490
- [Background] Berkley S, Chan M, Elias C, Fauci A, Lake A, Phumaphi J. Decade of Vaccines. Foreword. Vaccine. 2013 Apr 18;31 Suppl 2:B1-2. doi: 10.1016/j.vaccine.2013.02.014. No abstract available. PMID 23598469
- [Background] The World Bank. Information and communications for development 2012: Maximizing mobile. Washington, DC: The World Bank; 2012.
- [Background] Hayes, R.J. and Moulton, L.H. Clustered Randomised Trials. 2009, Chapman & Hall/CRC Press.
- [Result] Stockwell MS, Kharbanda EO, Martinez RA, Vargas CY, Vawdrey DK, Camargo S. Effect of a text messaging intervention on influenza vaccination in an urban, low-income pediatric and adolescent population: a randomized controlled trial. JAMA. 2012 Apr 25;307(16):1702-8. doi: 10.1001/jama.2012.502. PMID 22535855
- [Result] Stockwell MS, Westhoff C, Kharbanda EO, Vargas CY, Camargo S, Vawdrey DK, Castano PM. Influenza vaccine text message reminders for urban, low-income pregnant women: a randomized controlled trial. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):e7-12. doi: 10.2105/AJPH.2013.301620. Epub 2013 Dec 19. PMID 24354839
- [Result] Banerjee AV, Duflo E, Glennerster R, Kothari D. Improving immunisation coverage in rural India: clustered randomised controlled evaluation of immunisation campaigns with and without incentives. BMJ. 2010 May 17;340:c2220. doi: 10.1136/bmj.c2220. PMID 20478960
- [Result] Gebresilassie FE, Mariam DH. Factors influencing people's willingness-to-buy insecticide-treated bednets in Arbaminch Zuria District, southern Ethiopia. J Health Popul Nutr. 2011 Jun;29(3):200-6. doi: 10.3329/jhpn.v29i3.7867. PMID 21766555
- [Result] Bangure D, Chirundu D, Gombe N, Marufu T, Mandozana G, Tshimanga M, Takundwa L. Effectiveness of short message services reminder on childhood immunization programme in Kadoma, Zimbabwe - a randomized controlled trial, 2013. BMC Public Health. 2015 Feb 12;15:137. doi: 10.1186/s12889-015-1470-6. PMID 25885862